CLINICAL TRIAL: NCT06106685
Title: Washed Microbiota Transplantation for Chronic Constipation in Adults: a Single-center, Randomized, Double-blind, Placebo-controlled, Dose-exploring Clinical Study
Brief Title: Washed Microbiota Transplantation for Chronic Constipation in Adults
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The Second Hospital of Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: WMT-001-IIT-CC
Record Dates: First submitted 2023-10-12; First posted 2023-10-30 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-07

CONDITIONS: Constipation
Keywords: washed microbiota transplantation; constipation; difficult defecation
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- High-dose group (Experimental): The participant will receive a high dose of the washed microbiota suspension, with a bacterial quantity that is 10 times higher than the conventional clinical treatment dose, once daily for a duration of 4 days.
  Interventions: Drug: High-dose washed microbiota suspension
- Low-dose group (Experimental): The participant will receive a low-dose washed microbiota suspension, with a bacterial quantity equivalent to the conventional clinical treatment dose. The washed microbiota suspension will be administered once on the first day, followed by placebo of equal volume for the next 3 days.
  Interventions: Drug: Low-dose washed microbiota suspension
- Control group (Placebo Comparator): The patient will receive a placebo of equal volume once daily for a duration of 4 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: High-dose washed microbiota suspension — The high-dose group will be administered a high dose of washed microbiota suspension。
  Other Names: WMT-001
  Arms: High-dose group
Drug: Low-dose washed microbiota suspension — The low-dose group will be administered a low dose of washed microbiota suspension.
  Arms: Low-dose group
Drug: Placebo — The control group will be given equal volume placebo (120ml carrier solution matching the volume of WMT-001), which contains 10% sterile glycerol and saline injection. The drug was administered once a day for 4 days.
  Arms: Control group

SUMMARY:
This is a single-center, randomized, double-blind, placebo-controlled, dose-exploring clinical study to explore the safety and efficacy of washed microbiota transplantation (WMT) for patients with chronic constipation.

DETAILED DESCRIPTION:
At least 18 subjects who meet all the inclusion criteria but do not meet any exclusion criteria will be enrolled in this study. They will be randomly assigned to the high-dose group (high dose of washed microbiota suspension), the low-dose group (low dose of washed microbiota suspension) and the control group (placebo). Data of demographic characteristics, intestinal symptoms，medicine treatment usage and clinical outcomes will be collected. After treatment (D1-D4), they will enter the double-blind visit (D5, D18) for safety and efficacy evaluation. Open follow-up periods will be performed on days 32 and 60 after administration.

ELIGIBILITY:
Inclusion Criteria:

-

Meet all of the following inclusion criteria :

1. Voluntary sign informed consent, age 18-70 years old (including the threshold), male and female.
2. For subjects diagnosed with chronic constipation, the duration of the disease is at least 6 months, and the following conditions are met:

   1. Frequency of spontaneous defecation <3 times/week (spontaneous defecation refers to spontaneous defecation without the aid of remedial purgatives or manual assistance).
   2. Dry and hard stool: More than a quarter of the stool is type 1 or 2 on the Bristol Fecal Trait Scale.
3. The subject or his/her legal representative has given informed consent, is fully aware of the purpose of the study, is able to communicate well with the investigator, and is able to understand and comply with the requirements of the study.

Exclusion Criteria:

-

All exclusion criteria below are not met:

1. Outlet obstruction constipation, such as rectal mucosal prolapse.
2. History of abdominal and pelvic surgery, except for no intestinal complications after cholecystectomy, caesarean section, appendectomy, and treatment of intestinal polyps.
3. Combined with the colonoscopy results in the past 24 months, patients with intestinal stenosis caused by organic lesions of the digestive tract (such as tumor, inflammation, anal fissure, Crohn's disease, intestinal adhesion, ulcerative colitis, intestinal tuberculosis, etc.) and constipation.
4. Other systemic diseases involving the digestive tract (such as neurological diseases (such as Parkinson's disease, spinal cord injury, multiple sclerosis, etc.), muscle diseases (such as amyloidosis, dermatomyositis, etc.), mental disorders (such as depression, etc.), metabolic endocrine disorders (such as diabetes, hypothyroidism, etc.), or constipation caused by opioids.
5. Have a history of major surgery or severe trauma within 3 months and have not fully recovered.
6. There are contraindications for endoscopic intestinal catheterization via colonic approach, such as severe intestinal stenosis, obstruction, deep ulcer, and high risk of perforation. There are serious ulcers or a large number of false polyps in the fixation area, which is not suitable for fixation. The subject's behavior is seriously out of control.
7. Cardiac function and cardiac performance have any of the following abnormalities:

   1. According to the New York Heart Association (NYHA) heart function rating, the heart function rating is grade III and above.
   2. Subjects with new myocardial infarction or unstable angina pectoris within 6 months.
   3. Electrocardiogram indicated prolonged corrected QT interval (QTc) (male QTc≥450ms, female QTc≥470ms).
   4. Atrial arrhythmias that cannot be stably controlled by drugs and ventricular arrhythmias that require drug control (including grade 2 and above atrioventricular block).
8. Poor lung function that the investigator assessed as having an impact on study treatment, such as in subjects with acute chronic obstructive pulmonary disease or long-term oral, intravenous hormone control (other than inhalant/spray hormone use).
9. Uncontrolled immune disease and/or the need for long-term use of hormones (except for topical use).
10. Subjects with poorly controlled metabolic disease (e.g., thyroid dysfunction) or metabolic disease with gastrointestinal complications (e.g., gastrointestinal autonomic dysfunction, diabetic gastroparesis, etc.);
11. Patients with reproductive system diseases (including but not limited to ovarian cysts, endometriosis, primary dysmenorrhea, etc.) that are prone to abdominal pain.
12. Significant abnormalities in laboratory tests that, in the investigator's judgment, may affect subject safety or completion of the clinical study include:

    1. Hemoglobin <100g/L.
    2. Serum creatinine ≥1.5 times the upper limit of normal (ULN)
    3. Abnormal liver function, defined as Glutamic oxalacetic transaminase >1.5×ULN and/or Glutamic-pyruvic transaminase>1.5×ULN and/or total bilirubin >1.5×ULN.
    4. Coagulation function: PLT≤80×109/L, activated partial thromboplastin time > 1.5×ULN, prothrombin time > 1.5×ULN, International Normalized Ratio > 1.5×ULN.
    5. The results of routine stool or fecal occult blood are abnormal and have clinical significance to indicate gastrointestinal disease.
13. Subjects with active hepatitis who require or are on long-term use of therapeutic drugs, HIV, or active tuberculosis.
14. Subjects with a history of drug or alcohol abuse (i.e., consuming more than 14 servings (1 serving is 360mL) of beer, 45mL of 40% spirits, or 150mL of wine per week) or substance abuse.
15. Known allergy to the investigational drug, similar drugs or excipients.
16. Anti-infective drugs (antibiotics, antifungal, antiviral) were used within 14 days prior to enrollment, or anti-infective therapy was required at the time of enrollment evaluation.
17. Drugs and supplements that affect gastrointestinal motility and function that cannot be discontinued in trials, including but not limited to: antibiotics, such as erythromycin; Drugs that regulate intestinal microecology, such as probiotics such as Bifidobacterium; Parasympathetic inhibitors, such as scopolamine, atropine, belladonna, etc. Muscle relaxants such as succinylcholine; Antidiarrheal agents such as loperamide, Smecta, etc. Opioid preparations; Inhibition of gastric acid secretion drugs.
18. Those who use hydrotherapy for defecation/bowel cleansing within one month prior to treatment.
19. Women who are pregnant or breastfeeding, or who refuse to use effective contraception within 3 months after the last dose of medication.
20. Participants who had participated in clinical trials of drug intervention within 3 months before drug administration.
21. Patients with malignant tumors.
22. There are other situations in which the investigator deems it inappropriate to participate in this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2023-07-24 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
The incidence of treatment-related adverse events (AE) assessed by CTCAE, Version 5.0 | Two-week post-WMT
  The severity of AE was graded as mild (grade 1), moderate (grade 2), severe/disabling (grade 3), life threatening (grade 4), and death (grade 5). All AE were divided in definitely, probably and possibly related to treatment. The treatment-related AE we focused on included microbiota-related AEs (e.g., infection, diarrhea, abdominal pain, etc.) and route of delivery related AEs (e.g., nausea, vomiting, etc.).

SECONDARY OUTCOMES:
The incidence of treatment-related adverse events (AE) assessed by CTCAE, Version 5.0 | Day 5，Four-week post-WMT，Eight-week post-WMT
  The severity of AE was graded as mild (grade 1), moderate (grade 2), severe/disabling (grade 3), life threatening (grade 4), and death (grade 5). All AE were divided in definitely, probably and possibly related to treatment. The treatment-related AE we focused on included microbiota-related AEs (e.g., infection, diarrhea, abdominal pain, etc.) and route of delivery related AEs (e.g., nausea, vomiting, etc.).
The clinical response rate after treatment | One-week post-WMT，two-week post-WMT，Four-week post-WMT，Eight-week post-WMT
  A clinical response was defined as a patient achieving complete spontaneous bowel movement (CSBM) at least 50% of the time after receiving WMT. CSBM was defined as the number of spontaneous defecation with complete exhaust feeling without taking remedial purgative or manual assistance.
The weekly usage rate of assisted defecation drugs. | One-week post-WMT，Two-week post-WMT, Four-week post-WMT，Eight-week post-WMT
  Percentage of days per week after WMT that assisted defecation drugs were used, which was compared to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Faming Zhang, Principal Investigator — The Second Hospital of Nanjing Medical University
Locations (2):
- China (2):
  - The second affiliated hospital of Nanjing Medical University, Nanjing, Jiangsu
  - the Second Affiliated of Nanjing Medical University, Nanjing, Jiangsu

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pare P, Ferrazzi S, Thompson WG, Irvine EJ, Rance L. An epidemiological survey of constipation in canada: definitions, rates, demographics, and predictors of health care seeking. Am J Gastroenterol. 2001 Nov;96(11):3130-7. doi: 10.1111/j.1572-0241.2001.05259.x. PMID 11721760
- [Result] Long Y, Huang Z, Deng Y, Chu H, Zheng X, Yang J, Zhu Y, Fried M, Fox M, Dai N. Prevalence and risk factors for functional bowel disorders in South China: a population based study using the Rome III criteria. Neurogastroenterol Motil. 2017 Jan;29(1). doi: 10.1111/nmo.12897. Epub 2016 Jul 14. PMID 27412422
- [Result] Zhao YF, Ma XQ, Wang R, Yan XY, Li ZS, Zou DW, He J. Epidemiology of functional constipation and comparison with constipation-predominant irritable bowel syndrome: the Systematic Investigation of Gastrointestinal Diseases in China (SILC). Aliment Pharmacol Ther. 2011 Oct;34(8):1020-9. doi: 10.1111/j.1365-2036.2011.04809.x. Epub 2011 Aug 17. PMID 21848795
- [Result] Fleming V, Wade WE. A review of laxative therapies for treatment of chronic constipation in older adults. Am J Geriatr Pharmacother. 2010 Dec;8(6):514-50. doi: 10.1016/S1543-5946(10)80003-0. PMID 21356503
- [Result] Gallegos-Orozco JF, Foxx-Orenstein AE, Sterler SM, Stoa JM. Chronic constipation in the elderly. Am J Gastroenterol. 2012 Jan;107(1):18-25; quiz 26. doi: 10.1038/ajg.2011.349. Epub 2011 Oct 11. PMID 21989145
- [Result] Vazquez Roque M, Bouras EP. Epidemiology and management of chronic constipation in elderly patients. Clin Interv Aging. 2015 Jun 2;10:919-30. doi: 10.2147/CIA.S54304. eCollection 2015. PMID 26082622
- [Result] Mohaghegh Shalmani H, Soori H, Khoshkrood Mansoori B, Vahedi M, Moghimi-Dehkordi B, Pourhoseingholi MA, Norouzinia M, Zali MR. Direct and indirect medical costs of functional constipation: a population-based study. Int J Colorectal Dis. 2011 Apr;26(4):515-22. doi: 10.1007/s00384-010-1077-4. Epub 2010 Oct 19. PMID 20957375
- [Result] Lee-Robichaud H, Thomas K, Morgan J, Nelson RL. Lactulose versus Polyethylene Glycol for Chronic Constipation. Cochrane Database Syst Rev. 2010 Jul 7;(7):CD007570. doi: 10.1002/14651858.CD007570.pub2. PMID 20614462
- [Result] Chang L, Lacy BE, Moshiree B, Kassebaum A, Abel JL, Hanlon J, Bartolini W, Boinpally R, Bochenek W, Fox SM, Mallick M, Tripp K, Omniewski N, Shea E, Borgstein N. Efficacy of Linaclotide in Reducing Abdominal Symptoms of Bloating, Discomfort, and Pain: A Phase 3B Trial Using a Novel Abdominal Scoring System. Am J Gastroenterol. 2021 Sep 1;116(9):1929-1937. doi: 10.14309/ajg.0000000000001334. PMID 34465695
- [Result] Chey WD, Sayuk GS, Bartolini W, Reasner DS, Fox SM, Bochenek W, Boinpally R, Shea E, Tripp K, Borgstein N. Randomized Trial of 2 Delayed-Release Formulations of Linaclotide in Patients With Irritable Bowel Syndrome With Constipation. Am J Gastroenterol. 2021 Feb 1;116(2):354-361. doi: 10.14309/ajg.0000000000000967. PMID 33065589
- [Result] Zhang T, Lu G, Zhao Z, Liu Y, Shen Q, Li P, Chen Y, Yin H, Wang H, Marcella C, Cui B, Cheng L, Ji G, Zhang F. Washed microbiota transplantation vs. manual fecal microbiota transplantation: clinical findings, animal studies and in vitro screening. Protein Cell. 2020 Apr;11(4):251-266. doi: 10.1007/s13238-019-00684-8. Epub 2020 Jan 9. PMID 31919742
- [Result] Waitzberg DL, Logullo LC, Bittencourt AF, Torrinhas RS, Shiroma GM, Paulino NP, Teixeira-da-Silva ML. Effect of synbiotic in constipated adult women - a randomized, double-blind, placebo-controlled study of clinical response. Clin Nutr. 2013 Feb;32(1):27-33. doi: 10.1016/j.clnu.2012.08.010. Epub 2012 Aug 23. PMID 22959620
- [Result] Schoenfeld P, Lacy BE, Chey WD, Lembo AJ, Kurtz CB, Reasner DS, Bochenek W, Tripp K, Currie MG, Fox SM, Blakesley RE, O'Dea CR, Omniewski ND, Hall ML. Low-Dose Linaclotide (72 mug) for Chronic Idiopathic Constipation: A 12-Week, Randomized, Double-Blind, Placebo-Controlled Trial. Am J Gastroenterol. 2018 Jan;113(1):105-114. doi: 10.1038/ajg.2017.230. Epub 2017 Aug 22. PMID 29091082